CLINICAL TRIAL: NCT04049942
Title: The Comparison of a Short Home-based Multimodal Prehabilitation Strategy to Preoperative Aerobic Training Program on the Perioperative Functional Capacity and Outcomes in Patients Undergoing Thoracoscopic Lobectomy
Brief Title: Comparing the Impact of Multimodal Prehabilitation to Aerobic Training on Patients Undergoing Thoracoscopic Lobectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LZJ002
Record Dates: First submitted 2019-07-30; First posted 2019-08-08 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-08

CONDITIONS: Perioperative; Recovery; Prehabilitation; Thoracoschisis; Lobectomy; Lung Cancer
Keywords: Perioperative; Functional capability; Prehabilitation; Thoracoscopic lobectomy; Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation group (Experimental): Multimodal prehabilitation strategy includes physical exercise (moderate aerobic exercise combined with resistance exercise and respiratory training ), nutritional suggestion and optimization(whey protein supplement), and psychological therapy, as well as conventional guidance (including preoperative anesthesia assessment, drug treatment recommendations for chronic disease, quit smoking and abstinence). Patients are advised to record daily exercises and adherence to nutritional, psychological and other recommendations. Short message interviews are sent to patients twice a week to optimize adherence and promote feedback.
  Interventions: Other: Multimodal prehabilitation group
- Aerobic training group (Experimental): Aerobic training strategy includes the same guided individualized moderate aerobic exercise as the multimodal prehabilitation group, as well as the conventional guidance. Patients are advised to record daily exercises. Short message interviews are sent to patients twice a week to optimize adherence and promote feedback.
  Interventions: Behavioral: Aerobic training group

INTERVENTIONS:
Other: Multimodal prehabilitation group — Multimodal prehabilitation strategy includes physical exercise (moderate aerobic exercise combined with resistance exercise and respiratory training ), nutritional suggestion and optimization(whey protein supplement), and psychological therapy, as well as conventional guidance (including preoperative anesthesia assessment, drug treatment recommendations for chronic disease, quit smoking and abstinence). Patients are advised to record daily exercises and adherence to nutritional, psychological and other recommendations. Short message interviews are sent to patients twice a week to optimize adherence and promote feedback.
  Arms: Prehabilitation group
Behavioral: Aerobic training group — Aerobic training strategy includes the same guided individualized moderate aerobic exercise as the multimodal prehabilitation group, as well as the conventional guidance. Patients are advised to record daily exercises. Short message interviews are sent to patients twice a week to optimize adherence and promote feedback.
  Arms: Aerobic training group

SUMMARY:
In recent years, many studies have shown that prehabilitation based on aerobic training strategies could have a positive effect on the recovery of postoperative functional capacity in patients undergoing lung cancer surgery. Investigators are proposing a prospective randomized controlled trial to compare the impact of a short home-based multimodal prehabilitation strategy to preoperative aerobic training on patients scheduled for video-assisted thorascopic lobectomy for lung cancer. The multimodal prehabilitation strategy includes guided aerobic and resistance exercise, breathing exercises, nutrition supplement and physiology management preoperatively, while the aerobic strategy offers the same aerobic training guidance without the other parts. The prehabilitation lasts 2-3 weeks in our center. Investigators follow-up patients until 30 days after surgery, to investigate whether multimodal prehabilitation strategy differs from aerobic training program in postoperative functional capability improvement, health-related quality of life scorings, incidence of postoperative complications and other outcomes.

DETAILED DESCRIPTION:
This is a randomized controlled trial comparing the impact of a short home-based multimodal prehabilitaiton strategy to preoperative aerobic training program on patients undertaking video-assisted thoracoscopic (VATS) lobectomy for lung cancer.

The purpose of prehabilitation is to enhance an individual's functional capacity to reach the optimal physiological state before surgery, helping them withstand the stress of surgery and receive an enhanced recovery post operation. Recent studies have shown that trimodal or multimodal prehabilitation strategy including exercise, diet and psychologic guidance could improve postoperative functional recovery for patients undergoing colorectal resection. However, researches regarding to the effect of multi-modal prehabilitation in other types of operations remain scarce.

Studies have shown that the postoperative functional capacity decreases in patients undergoing lung cancer surgery. Therefore, many clinical trials were designed to explore the impact of prehabilitation on these patients, and many of them yielded positive results, showing preoperative exercise for patients undergoing lung cancer surgery is safe and beneficial in postoperative functional capacity recovery. However, the majority of the trials conducted adopted preoperative exercises, specifically aerobic exercises, as the sole means of prehabilitation. In 2017, our team conducted a randomized controlled trial (registration number NCT03068507) to examine the efficacy of a 2-week multimodal home-based prehabilitation strategy in patients undergoing VATS lobectomy for lung cancer. The preliminary results indicate that patients who received the short multimodal home-based prehabilitation have a significantly higher 6-minute walk distance (6MWD) perioperatively.

Investigators are proposing a new randomized controlled trial to compare the efficacy of a short multimodal home-based prehabilitation with the sole aerobic prehabilitation strategy adopted by the previous studies.

A total of 100 patients scheduled to have elective VATS lobectomy for primary lung cancer will be recruited in this research at Peking Union Medical College Hospital. After informed consent is obtained, the patients will be evenly assigned to two groups randomly based on computer-generated sequence, the multimodal prehabilitation group and the aerobic prehabilitation group. The random allocation will be concealed using sealed opaque envelops.

The multimodal group will receive an individualized prehabilitation strategy after a complete assessment, including aerobic and resistance exercise, nutritional optimization, and psychological therapy, as well as conventional guidance. All patients will receive an instruction booklet with details in text and pictures, and will be asked to complete standard diaries in the booklet. The length of prehabilitation will be 2-3 weeks, determined by the waiting time till surgery alone.

For the multimodal group, prehabilitation strategy is as follows: 1) a 30-minute aerobic exercise at least 3 times a week, in the form of jogging, power walking or cycling, according to the patients' individual choice; 2) a guided resistance exercise at least twice a week, using a pull strap distributed by investigators to accomplish 4 pre-set resistance posture; 3) breathing exercise at least 3 times per day, lasting over 10 minutes, in the form of guided effective coughing, blowing up a small balloon or using the respiratory exerciser distributed by investigators; 4) nutritional advice and whey protein supplement 1hour prior to exercising (20g/day for male and 15g/day for female patients); 5) psychological therapy by listening to soothing music or radio and other relaxing activities. Patients are advised to record daily exercises and adherence to nutritional, psychological and other recommendations in a prehabilitation journal distributed by investigators. Standardized short message interviews are sent to patients twice a week to optimize adherence and promote timely feedback.

The aerobic group will receive the same guidance in the individualized home-based aerobic exercise strategy as the multimodal group, but not in the other aspects. These patients are also advised to keep a prehabilitation journal recording daily exercises and will receive the same short message interviews twice a week.

All patients enrolled will receive the conventional guidance, including preoperative anesthesia assessment, drug treatment recommendations for chronic disease, quit smoking and abstinence. And patients are also provided some useful information about anesthesia and surgery process.

The patients and trial personnel will not be blinded to the allocation regarding to the nature of the intervention. The outcome assessors will independently collect the outcome data without the knowledge of the allocation.

The primary outcome will be post-operative 6-minute walk distance (6MWD), measured as functional walking capacity, at 30 days postoperatively). The secondary outcomes include perioperative 6MWD (1 day before surgery, 30 days postoperatively), pulmonary function (1 day before surgery, 30 days postoperatively), hospital anxiety and depression scale (HADS), World Health Organization disability assessment schedule II (WHODAS 2.0) score, postoperative quality of recovery score -15 (QoR-15) score and prognosis information (mortality and morbidity, length of hospital stay, ICU stay time, duration of chest tube, etc.).

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient of thoracic surgery department in Peking Union Medical College Hospital
2. From 18y/o to 70y/o
3. Suspected of lung cancer
4. Decide to take the elective thoracoscopic surgery in Peking Union Medical College Hospital

Exclusion Criteria:

1. Decline to participant the study (due to any reason)
2. American Society of Anesthesiologists (ASA) grade >III
3. TNM stage I-III
4. Patients plan to receive neoadjuvant therapy
5. Unable to tolerate prehabilitaion or aerobic strategy (including exercise guide, whey protein and psycho-relaxation exercise)
6. Other severe cardio-pulmonary diseases that would affect the 6MWD

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
post-operative 6-minute walk distance | 30 days postoperatively
  Use 6-minute walk distance (6MWD) to evaluate the physical functional capability objectively. The primary outcome will be analyzed after stratification by age and baseline functional capacity.

SECONDARY OUTCOMES:
Perioperative 6MWD | baseline, 1 day before surgery
  Evaluate the impact of prehabilitation on functional capability before surgery.
Perioperative pulmonary functional test | Baseline, 1 day before surgery, 30 days postoperatively
  Evaluate the recovery of pulmonary capacity. Forced expiratory volume in 1 s (FEV1) and forced vital capacity (FVC) will be measured in liters, and FEV1/FVC will be calculated with the FEV1 and FVC value and reported in percentage.
Perioperative Hospital Anxiety and Depression Scale (HADS) | Baseline, 1 day before surgery, 30 days postoperatively
  The HADS is a questionnaire composed of 14 questions to screen for anxiety and depression. The questionnaire features 7 questions on anxiety and seven on depression. The maximum score for either anxiety or depression is 21 and the minimum for either is 0. The severity of anxiety and depression correlates with the scoring. HADS will be used to evaluate the mental capability recovery after surgery.
WHO disability assessment schedule 2.0 (WHODAS 2.0) | Baseline, 1 day before surgery, 30 days postoperatively
  WHODAS 2.0 is a patient self-report assessment tool that evaluates the patient's ability to perform activities in six domains of functioning over the previous 30 days. Each item from the six domains is rated using a 5-point Likert scale (1 = no difficulty, 2 = mild difficulty, 3 = moderate difficulty, 4 = severe difficulty, 5 = extreme difficulty). These are then calculated to get a score representing global disability. WHODAS 2.0 will be adopted to make the the global evaluation of patients' disability before and after surgery.
Postoperative quality of recovery score -15 (QoR-15) | the 1st, 2nd and 3rd day postoperatively
  QoR-15 is an easy-to-use score for assessing the quality of post-operative recovery. It is a questionnaire featuring 15 items, each of which has a scale of 0 to 10. Higher scores of QoR-15 indicate better recovery quality after surgery. QoR-15 will be used in this study to evaluate the intermediate phase of recovery.
Prognosis information1: mortality | 30 days postoperatively
  Evaluate postoperative all-cause mortality, reported in percentage.
Prognosis information2: morbidity | 30 days postoperatively
  Evaluate the incidence of major postoperative complications including atelectasis, pneumonia, respiratory failure, sepsis, septic shock, which will be all reported in percentage.
Prognosis information3: length of hospital stay | 30 days postoperatively
  Evaluate postoperative length of hospital stay, reported in days.
Prognosis information4: ICU stay time | 30 days postoperatively
  Evaluate postoperative ICU stay time, reported in days.
Prognosis information5: duration of chest tube | 30 days postoperatively
  Evaluate duration of chest tube placement, reported in days.

CONTACTS AND LOCATIONS:
Overall Officials: Yuguang HUANG, M.D., Study Chair — Peking Union Medical College Hospital, Chinese Academy of Medicine Sciences
Locations (1):
- PekingUnionMedicalCollegeHospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Liu Y, Liu Z, Zhang Y, Cui Y, Pei L, Huang Y. The protocol for the prehabilitation for thoracic surgery study: a randomized pragmatic trial comparing a short home-based multimodal program to aerobic training in patients undergoing video-assisted thoracoscopic surgery lobectomy. Trials. 2023 Mar 15;24(1):194. doi: 10.1186/s13063-023-07220-4. PMID 36922827